CLINICAL TRIAL: NCT06108180
Title: Effectiveness of the Dry Needling Approach in Patients With Tension-Type Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Sofía Monti Ballano, Principal Investigator, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RAT 2023-195
Record Dates: First submitted 2023-10-20; First posted 2023-10-30 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Tension-Type Headache; Dry Needling
MeSH Terms: conditions — Tension-Type Headache | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry Needling group (Experimental)
  Interventions: Other: Dry Needling
- Control group (No Intervention)

INTERVENTIONS:
Other: Dry Needling — 3 treatment to eliminate active trigger points that patients have
  Arms: Dry Needling group

SUMMARY:
Randomized Single-Blind Clinical Trial in which the treatment will be administered through 3 sessions of dry needling in the cervical, cranial, and facial musculature in patients with frequent and chronic tension-type headache.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of tension headache according to IHS

Exclusion Criteria:

* Documented major trauma through medical history in the cervical area and/or recent surgery.
* Pregnancy.
* Generalized pain.
* Inflammatory, hormonal, or neurological disorders.
* Tendon disorders in the upper extremities.
* Severe psychiatric illnesses.
* Inability to complete the form in Spanish.
* Having a pacemaker (due to the use of equipment with magnetic sensors).
* Specific contraindications to invasive or conservative physiotherapy (infection, fever, hypothyroidism, wounds in the puncture area, metal allergies, cancer, systemic diseases, or belonephobia).
* Having received physiotherapy treatment for the condition in the past month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-10-23 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
Active trigger points | 1 month
  The investigators assess the sensitivity of trigger points using algometry to determine which points reproduce the participants tensional-type headache.

SECONDARY OUTCOMES:
cervical ROM | 1 month
  general cervical range of movement, upper and lower cervical

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Clínico de Fisioterapia OMT-E, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferrante T, Manzoni GC, Russo M, Camarda C, Taga A, Veronesi L, Pasquarella C, Sansebastiano G, Torelli P. Prevalence of tension-type headache in adult general population: the PACE study and review of the literature. Neurol Sci. 2013 May;34 Suppl 1:S137-8. doi: 10.1007/s10072-013-1370-4. PMID 23695063
- [Background] Fernandez-de-Las-Penas C, Ge HY, Arendt-Nielsen L, Cuadrado ML, Pareja JA. The local and referred pain from myofascial trigger points in the temporalis muscle contributes to pain profile in chronic tension-type headache. Clin J Pain. 2007 Nov-Dec;23(9):786-92. doi: 10.1097/AJP.0b013e318153496a. PMID 18075406
- [Background] Cerezo-Tellez E, Torres-Lacomba M, Fuentes-Gallardo I, Perez-Munoz M, Mayoral-Del-Moral O, Lluch-Girbes E, Prieto-Valiente L, Falla D. Effectiveness of dry needling for chronic nonspecific neck pain: a randomized, single-blinded, clinical trial. Pain. 2016 Sep;157(9):1905-1917. doi: 10.1097/j.pain.0000000000000591. PMID 27537209
- [Background] Stephens LR, Humphrey JD, Little PB, Barnum DA. Morphological, biochemical, antigenic, and cytochemical relationships among Haemophilus somnus, Haemophilus agni, Haemophilus haemoglobinophilus, Histophilus ovis, and Actinobacillus seminis. J Clin Microbiol. 1983 May;17(5):728-37. doi: 10.1128/jcm.17.5.728-737.1983. PMID 6408118